CLINICAL TRIAL: NCT02246179
Title: Fractional Carbon Dioxide Laser Assisted Delivery of Topical Anesthetics: a Randomized Controlled Pilot Study
Brief Title: Fractional Laser Assisted Delivery of Anesthetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NL48655.018.14
Record Dates: First submitted 2014-09-12; First posted 2014-09-22 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Local Anesthesia of the Skin.
Keywords: Fractional laser; Topical anesthesia; Drug delivery
MeSH Terms: interventions — Carticaine; Epinephrine; Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: AFXL + AHES (Experimental): This test region will be pretreated with a fractional carbon dioxide laser (ablative fractional laser; AFXL) with a 120 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse at t0 in a subject blinded fashion. Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will be applied at this test region at t1.Ten minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at t11 to the subject at the test region using AFXL at 5% density and 35 mJ/microbeam.
  Interventions: Device: AFXL; Drug: AHES
- 2: AFXL + EMLA (Experimental): This test region will be pretreated with a fractional carbon dioxide laser (ablative fractional laser; AFXL) with a 120 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse at t0 in a subject blinded fashion. Eutectic mixture of lidocaine 25 mg/g and prilocaine 25 mg/g cream (EMLA cream) will be applied at this test region at t1.Ten minutes after EMLA cream application (incubation time; under occlusion), a pain stimulus will be given at t11 to the subject at the test region using AFXL at 5% density and 35 mJ/microbeam.
  Interventions: Device: AFXL; Drug: EMLA cream
- 3: Sham AFXL + AHES (Sham Comparator): A pass with a fractional carbon dioxide laser with a 120 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse will be given at the area right adjacent to this test region ("sham AFXL") at t0 in a subject blinded fashion. Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will then be applied at this test region on the intact skin at t1. Ten minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at t11 to the subject at the test region using AFXL at 5% density and 35 mJ/microbeam.
  Interventions: Device: AFXL; Drug: AHES
- 4: Sham AFXL + EMLA (Sham Comparator): A pass with a fractional carbon dioxide laser with a 120 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam, single pulse will be given at the area right adjacent to this test region ("sham AFXL") at t0 in a subject blinded fashion. Eutectic mixture of lidocaine 25 mg/g and prilocaine 25 mg/g cream (EMLA cream) will then be applied at this test region on the intact skin at t1. Ten minutes after EMLA cream application (incubation time; under occlusion), a pain stimulus will be given at t11 to the subject at the test region using AFXL at 5% density and 35 mJ/microbeam.
  Interventions: Device: AFXL; Drug: EMLA cream

INTERVENTIONS:
Device: AFXL — Pretreatment at 2.5 mJ/microbeam and 5% density Pain stimulus at 35 mJ/microbeam and 5% density
  Other Names: Fractional carbon dioxide laser; Ablative fractional laser; Fractional CO2 laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.
Drug: AHES — Topical application at test region 1 and 3 under occlusion for 10 minutes
  Other Names: Ultracain D-S forte; articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml
  Arms: 1: AFXL + AHES; 3: Sham AFXL + AHES
Drug: EMLA cream — Topical application at test region 2 and 4 under occlusion for 10 minutes
  Other Names: lidocaine 25 mg/g + prilocaine 25 mg/g cream
  Arms: 2: AFXL + EMLA; 4: Sham AFXL + EMLA

SUMMARY:
The purpose of this study is to assess the efficacy of fractional CO2 laser assisted delivery of topically applied anesthetics (articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution and EMLA cream) regarding to anesthesia of the skin.

DETAILED DESCRIPTION:
Rationale: In dermatology, many minor surgical and laser procedures are carried out under local anesthesia of the skin. Anesthesia using topical formulations is time consuming, as the anesthetic has to be applied at least one hour before treatment, and is often only partially effective. On the other hand infiltration anesthesia is often associated with discomfort and is not tolerated by patients who are for example needle phobic. In the past years, enhanced and accelerated penetration of various topically applied substances, including photosensitizers, has been proven by pretreatment of the skin with a fractional laser, creating a pattern of microscopic ablation craters.(Haedersdal et al., 2010) This improvement in drug penetration seems to be regardless of ablation crater depth.(Haak et al., 2012) There is limited evidence that transdermal lidocaine absorption can be increased by fractional laser pretreatment.(Oni et al., 2012; Oni et al., 2013) These findings might suggest that local anesthesia of the skin may be achieved by applying an anesthetic drug topically on a skin surface pretreated with a fractional laser. However, little is known about the role of the formulation of the topical drug delivered using this method.

Objective: The primary objective of this study is to assess the analgesic effect of fractional carbon dioxide laser assisted delivery of two topical anesthetics (articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) and EMLA cream) compared to application of these anesthetics without fractional laser pretreatment. The secondary objective is to compare the efficacy of these two different anesthetics, when applied according to the fractional laser drug delivery principle.

Study design: Prospective, single blinded, randomized, controlled, within subject, pilot study.

Study population: 10 healthy volunteers ≥18 years, who give written informed consent Intervention: In each subject, four test regions on subject's back of 1x1 centimeter will be randomly allocated in a 2x2 design to (1) ablative fractional laser (AFXL) pretreatment (5% density, 2.5 mJ/microbeam) followed by topical application of AHES, (2) AFXL pretreatment followed by application of EMLA cream, (3) sham AFXL followed by application of AHES on the intact skin and (4) sham AFXL followed by application of EMLA cream on the intact skin. Sham AFXL will be done by delivering an AFXL pass at 5% density and 2.5 mJ/microbeam right adjacent to the region of AHES or EMLA application on the intact skin. After ten minutes incubation time, an AFXL pass will be given as a pain stimulus at each test region with 5% density and 35 mJ/microbeam. Subjects will be asked to indicate pain on a visual analogue scale (VAS) from 0-10 (0: no pain; 10: worst imaginable pain) directly after each pain stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I or II
* Age ≥18 years
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* History of keloid or hypertrophic scar formation or complicated wound healing
* Presence of any active skin disease
* Known allergy to local anesthesia
* Pregnancy or lactation
* Incompetency to understand what the procedure involves
* Current complaints of chronic pain or other alterations in pain sensation (e.g. due to diabetes mellitus or lepra)
* Current treatment with systemic analgesics or other medication that can influence pain sensation
* Current treatment with anticoagulants
* Fitzpatrick skin type III-VI
* Excessive sun tan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain score | Directly after pain stimulus. After 10 minutes incubation time of the anesthetics.
  The main study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain) directly after each pain stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD, PhD, Principal Investigator — Netherlands Institute for Pigment Disorders, Department of Dermatology, Academic Medical Center, University of Amsterdam; Menno A. De Rie, MD, PhD, Study Director — Department of Dermatology, Academic Medical Center, University of Amsterdam
Locations (1):
- Netherlands Institute for Pigment disorders, Amsterdam, Netherlands

REFERENCES:
- [Background] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Background] Haak CS, Farinelli WA, Tam J, Doukas AG, Anderson RR, Haedersdal M. Fractional laser-assisted delivery of methyl aminolevulinate: Impact of laser channel depth and incubation time. Lasers Surg Med. 2012 Dec;44(10):787-95. doi: 10.1002/lsm.22102. Epub 2012 Dec 4. PMID 23212624
- [Background] Oni G, Brown SA, Kenkel JM. Can fractional lasers enhance transdermal absorption of topical lidocaine in an in vivo animal model? Lasers Surg Med. 2012 Feb;44(2):168-74. doi: 10.1002/lsm.21130. Epub 2012 Feb 2. PMID 22302761
- [Background] Oni G, Rasko Y, Kenkel J. Topical lidocaine enhanced by laser pretreatment: a safe and effective method of analgesia for facial rejuvenation. Aesthet Surg J. 2013 Aug 1;33(6):854-61. doi: 10.1177/1090820X13496248. PMID 23908302
- [Background] Ong MW, Bashir SJ. Fractional laser resurfacing for acne scars: a review. Br J Dermatol. 2012 Jun;166(6):1160-9. doi: 10.1111/j.1365-2133.2012.10870.x. Epub 2012 May 8. PMID 22296284
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] Hahn IH, Hoffman RS, Nelson LS. EMLA-induced methemoglobinemia and systemic topical anesthetic toxicity. J Emerg Med. 2004 Jan;26(1):85-8. doi: 10.1016/j.jemermed.2003.03.003. PMID 14751483
- [Background] Baron ED, Harris L, Redpath WS, Shapiro H, Hetzel F, Morley G, Bar-Or D, Stevens SR. Laser-assisted penetration of topical anesthetic in adults. Arch Dermatol. 2003 Oct;139(10):1288-90. doi: 10.1001/archderm.139.10.1288. PMID 14568832
- [Background] Koh JL, Harrison D, Swanson V, Norvell DC, Coomber DC. A comparison of laser-assisted drug delivery at two output energies for enhancing the delivery of topically applied LMX-4 cream prior to venipuncture. Anesth Analg. 2007 Apr;104(4):847-9. doi: 10.1213/01.ane.0000257925.36641.9e. PMID 17377092
- [Background] Shapiro H, Harris L, Hetzel FW, Bar-Or D. Laser assisted delivery of topical anesthesia for intramuscular needle insertion in adults. Lasers Surg Med. 2002;31(4):252-6. doi: 10.1002/lsm.10101. PMID 12355570
- [Background] Hantash BM, Bedi VP, Chan KF, Zachary CB. Ex vivo histological characterization of a novel ablative fractional resurfacing device. Lasers Surg Med. 2007 Feb;39(2):87-95. doi: 10.1002/lsm.20405. PMID 17115384
- [Background] Haak CS, Bhayana B, Farinelli WA, Anderson RR, Haedersdal M. The impact of treatment density and molecular weight for fractional laser-assisted drug delivery. J Control Release. 2012 Nov 10;163(3):335-41. doi: 10.1016/j.jconrel.2012.09.008. Epub 2012 Sep 21. PMID 23000695
- [Background] Togsverd-Bo K, Haak CS, Thaysen-Petersen D, Wulf HC, Anderson RR, Haedersdal M. Intensified photodynamic therapy of actinic keratoses with fractional CO2 laser: a randomized clinical trial. Br J Dermatol. 2012 Jun;166(6):1262-9. doi: 10.1111/j.1365-2133.2012.10893.x. PMID 22348388